CLINICAL TRIAL: NCT05922865
Title: Tri-service General Hospital, National Defence Medical Center, Taipei, Taiwan
Brief Title: The Effect of Smart Sensor Combined With APP for Individualized Precise Exercise Training in Long Covid-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shang-Lin Chiang (Other)
Responsible Party: Sponsor-Investigator, Shang-Lin Chiang, Attending physician, National Defense Medical Center, Taiwan
Organization: National Defense Medical Center, Taiwan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: smart knee assistive device
Record Dates: First submitted 2023-06-26; First posted 2023-06-28 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Coronavirus Disease; COVID-19; Long Covid-19; Telerehabilitation
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KNEESUP smart knee assistive device + KNEESUP care APP (Experimental): The participants with KNEESUP smart knee assistive device and KNEESUP care APP do exercise training at home.
  Interventions: Device: KNEESUP smart knee assistive device + KNEESUP care APP
- Health consultation (Placebo Comparator): The participants with healthy consultation do exercise training at home.
  Interventions: Behavioral: Healthy consulation

INTERVENTIONS:
Device: KNEESUP smart knee assistive device + KNEESUP care APP — In KNEESUP smart knee assistive device + KNEESUP care APP group, participants used the KNEESUP intelligent knee assistive device. Participants wore a knee brace with a sensor module on one side of the leg, the sensor could connect with the KNEESUP care APP which were installed in participant's mobile phone. The APP was designed with an individualized exercise program and the knee brace sensor could detect the action moment of the participants during exercise. This equipment could help the participants to achieve professional-level home rehabilitation.
  Arms: KNEESUP smart knee assistive device + KNEESUP care APP
Behavioral: Healthy consulation — In Healthy consulation group, participants received routine outpatient health education.
  Arms: Health consultation

SUMMARY:
The coronavirus (COVID -19) has rapidly turned into a global pandemic. For patients diagnosed with COVID-19, it caused severe damage in the upper respiratory system and systemic complications, including the cardiovascular, mental, nervous, and musculoskeletal system. Previous research has indicated that these subsequent sequelae can reduce quality of life. (A. W. Wong et al., 2020) Studies have indicated that exercise training is beneficial to improve blood pressure, reduce cardiovascular factors, reduce complications, and relieve depression (J. Galloza et al., 2017) However, the current international research on the benefits of exercise rehabilitation and the improvement of quality of life in patients who have been infected with COVID-19 is still lacking. Under the international epidemic, it is pointed out that the importance of telerehabilitation has also been advocated worldwide. Previous systematic review indicated that no matter it is nervous, muscular or cardiac system disease, the efficacy of telerehabilitation is superior to face-to-face rehabilitation. The purpose of this study is to compare the effect between the intervention of KNEESUP smart knee assistive device, and the health education in routine outpatient after diagnosis of Long Covid-19.

DETAILED DESCRIPTION:
The purpose of KNEESUP measuring equipment used in this research is to improve the recovery rate and reduce the sequelae after treatment. KNEESUP connects the subjects and researchers through technologies such as IoT and AI. The evaluation of the rehabilitation results can be presented as a data chart, and the treatment effects are also clearly presented.

For the subject, the subject puts on KNEESUP knee pads in a long sitting position, bends the knees about 30 degrees, aligns the position of the knee pad circle with the bone, and uses the strap on the lower side, upper side, and the knee pads. After wearing, press and hold the sensor on the outer side of the knee pad for 3 seconds, and then open the mobile app. After the hardware setting and connection are completed, the evaluation and exercise can begin.

ELIGIBILITY:
Inclusion Criteria:

* symptoms last at least one month after recovery
* without physical impairment
* understood verbal or non-verbal communication
* normal cognitive function
* were willing to participate in the study and accept random allocation

Exclusion Criteria:

* diagnosed with transient ischemic attack or stroke
* had neuromuscular injury or surgery in the lower limbs in the past six months
* had heart rhythm regulator
* hospitalized during training
* had aggravated symptoms due to infection again
* had participated in other clinical trials or received other alternative treatments

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Aerobic capacity (VO2 max in ml/kg/min ) | baseline, 12 weeks
  Maximal VO2 during testing, also means aerobic capacity
Anaerobic Threshold (mL/kg/min) | baseline, 12 weeks
  Anaerobic Threshold (AT) refers to the exercise intensity at which lactate begins to accumulate in the blood at a faster rate than it can be removed. It represents a transition point between predominantly aerobic metabolism (using oxygen) and increased anaerobic metabolism (without sufficient oxygen).
Working load in watt | baseline, 12 weeks
  Maximal Working load during testing
Breathing reserve (ml/kg/min) | baseline, 12 weeks
  A measure used during cardiopulmonary exercise testing (CPET) to assess how much of a person's maximum ventilatory capacity is unused at peak exercise. It reflects the difference between the maximum voluntary ventilation (MVV) and the minute ventilation (VE) reached during exercise.
Rest Heart rate in beat/min | baseline, 12 weeks
  Resting heart rate during exercise testing
O2 pulse in ml/beat | baseline, 12 weeks
  It means the heart pumps O2 volume by each heart beat, and also means left ventricle function.
Systolic blood pressure in mm Hg | baseline, 12 weeks
  The resting blood pressure during exercise testing
Diastolic blood pressure in mm Hg | baseline, 12 weeks
  The resting blood pressure during exercise testing
VE/VCO2 slope | baseline, 12 weeks
  The ventilation/ perfusion abnormalities (VE/VCO2) is measured by graded exercise testing.The change in VE/VCO2 was calculated as the value at 12 weeks minus the value at baseline. A lower VE/VCO2 ratio indicates better ventilatory efficiency and reduced ventilation/perfusion abnormalities.
Heart rate recovery | baseline, 12 weeks
  The heart rate recovery is measured by graded exercise testing, including 1 minute and 2 minute recovery.
  The change in heart rate recovery was calculated as the difference between heart rate recovery at 12 weeks and heart rate recovery at baseline. A decrease of < 12 or 22 beats per minute in 1- or 2- min heart rate recovery, respectively, indicates an elevated risk of mortality. A faster heart rate recovery indicates better cardiovascular fitness and autonomic regulation.
FVC (L/min) | baseline, 12 weeks
  The total amount of air exhaled (mL) during a forced expiratory volume test will be measured by spirometry. The change in FVC was calculated as the value at 12 weeks minus the value at baseline. A higher FVC indicates better lung function.
FEV1 (L/min) | baseline, 12 weeks
  The amount of air exhaled (mL) during the first second during a forced expiratory volume test will be measured by spirometry. The change in FEV1 was calculated as the value at 12 weeks minus the value at baseline. A higher FEV1 indicates better lung function.
FEV1/FVC (%) | baseline, 12 weeks
  The measured FEV1 is divided by the measured FVC. he change in FEV1/FVC was calculated as the value at 12 weeks minus the value at baseline. A higher FEV1/FVC ratio generally indicates better lung function, while a lower ratio suggests airflow limitation.
Gait: Step length (m) through Time Up and Go Test | baseline, 12 weeks
  Analysis software was evaluated using METASENS. Begin by having the participants sit back in a standard arm chair and identify a 3 meters line on the floor. Participants walk forward three meters at the usual speed, turn around and return to the chair before sitting down. The METASENS evaluation analysis software calculates the step length (m), speed (m/s), cadence (steps per minute), left/right gait cycle (sec), left/right knee flexion angle (deg), left/right foot contact extension angle (deg), turn around time (sec), stand up time (sec), total walking time (sec).
Gait: Speed (m/s) through Time Up and Go Test | baseline, 12 weeks
  Analysis software was evaluated using METASENS. Begin by having the participants sit back in a standard arm chair and identify a 3 meters line on the floor. Participants walk forward three meters at the usual speed, turn around and return to the chair before sitting down. The METASENS evaluation analysis software calculates the step length (m), speed (m/s), cadence (steps per minute), left/right gait cycle (sec), left/right knee flexion angle (deg), left/right foot contact extension angle (deg), turn around time (sec), stand up time (sec), total walking time (sec).
Gait: Cadence (steps per minute) through Time Up and Go Test | baseline, 12 weeks
  Analysis software was evaluated using METASENS. Begin by having the participants sit back in a standard arm chair and identify a 3 meters line on the floor. Participants walk forward three meters at the usual speed, turn around and return to the chair before sitting down. The METASENS evaluation analysis software calculates the step length (m), speed (m/s), cadence (steps per minute), left/right gait cycle (sec), left/right knee flexion angle (deg), left/right foot contact extension angle (deg), turn around time (sec), stand up time (sec), total walking time (sec).
Gait: Left gait cycle (sec) through Time Up and Go Test | baseline, 12 weeks
  Analysis software was evaluated using METASENS. Begin by having the participants sit back in a standard arm chair and identify a 3 meters line on the floor. Participants walk forward three meters at the usual speed, turn around and return to the chair before sitting down. The METASENS evaluation analysis software calculates the step length (m), speed (m/s), cadence (steps per minute), left/right gait cycle (sec), left/right knee flexion angle (deg), left/right foot contact extension angle (deg), turn around time (sec), stand up time (sec), total walking time (sec).
Gait: Right gait cycle (sec) through Time Up and Go Test | baseline, 12 weeks
  Analysis software was evaluated using METASENS. Begin by having the participants sit back in a standard arm chair and identify a 3 meters line on the floor. Participants walk forward three meters at the usual speed, turn around and return to the chair before sitting down. The METASENS evaluation analysis software calculates the step length (m), speed (m/s), cadence (steps per minute), left/right gait cycle (sec), left/right knee flexion angle (deg), left/right foot contact extension angle (deg), turn around time (sec), stand up time (sec), total walking time (sec).
Gait: Turn around time (sec) through Time Up and Go Test | baseline, 12 weeks
  Analysis software was evaluated using METASENS. Begin by having the participants sit back in a standard arm chair and identify a 3 meters line on the floor. Participants walk forward three meters at the usual speed, turn around and return to the chair before sitting down. The METASENS evaluation analysis software calculates the step length (m), speed (m/s), cadence (steps per minute), left/right gait cycle (sec), left/right knee flexion angle (deg), left/right foot contact extension angle (deg), turn around time (sec), stand up time (sec), total walking time (sec).
Gait: Stand up time (sec) through Time Up and Go Test | baseline, 12 weeks
  Analysis software was evaluated using METASENS. Begin by having the participants sit back in a standard arm chair and identify a 3 meters line on the floor. Participants walk forward three meters at the usual speed, turn around and return to the chair before sitting down. The METASENS evaluation analysis software calculates the step length (m), speed (m/s), cadence (steps per minute), left/right gait cycle (sec), left/right knee flexion angle (deg), left/right foot contact extension angle (deg), turn around time (sec), stand up time (sec), total walking time (sec).
Gait: Total walking time (sec) through Time Up and Go Test | baseline, 12 weeks
  Analysis software was evaluated using METASENS. Begin by having the participants sit back in a standard arm chair and identify a 3 meters line on the floor. Participants walk forward three meters at the usual speed, turn around and return to the chair before sitting down. The METASENS evaluation analysis software calculates the step length (m), speed (m/s), cadence (steps per minute), left/right gait cycle (sec), left/right knee flexion angle (deg), left/right foot contact extension angle (deg), turn around time (sec), stand up time (sec), total walking time (sec).
Long COVID symptoms | baseline, 12 weeks
  A simple checklist to record Long COVID symptoms. Symptoms that persisted or were newly developed after acute infection were documented as sequelae. Symptoms included fatigue, shortness of breath, cognitive dysfunction (referred to as "brain fog"), chest pain, cough, dizziness, headache, sleep disturbances, palpitations, depression/anxiety, and olfactory dysfunction.

SECONDARY OUTCOMES:
Quality of life (scores) | baseline, 12 weeks
  The Taiwanese version of the WHO Quality of Life-BREF (WHOQOL-BREF) with good validity and reliability includes the globally standardized WHOQOL-BREF with 26 items and an additional two locally developed items, making a total of 28 items. It consists of two single-facet items measuring overall quality of life and general health and four domains, including physical (7 items), psychological (6 items), social (4 items), and environmental (9 items) domains. The two additional items are being respected/accepted facet in the social domain and eating/food facet in the environment domain, respectively. The participants rated all items on a scale of 1-5, with higher scores reflecting a greater quality of life. Domain scores were derived by multiplying the mean of the facet scores within each domain by a scaling factor of 4, resulting in potential domain scores ranging from 4 to 20.
Sleeping Quality (scores) | baseline, 12 weeks
  Symptoms of sleeping quality will be assessed using Pittsburgh Sleeping Index. The content is aimed at the sleep conditions of the subjects, including seven items including personal self-evaluation of sleep quality, sleep latency, sleep hours, sleep efficiency, sleep disturbance, drug use and daytime dysfunction. Each item is calculated by the Likert four-point method, 0-3 points, the total score ranges from 0-21 points, and the higher the score, the worse the sleep quality. (MORGAN, DALLOSSO, EBRAHIM, ARIE, & Fentem, 1988; Tang Zhenqing et al., 2014).
Body composition: Body weight (kg) | baseline, 12 weeks
  The InBody device is a bioelectrical impedance analysis (BIA) system designed to assess body composition in a non-invasive, rapid, and reliable manner. It quantifies key components such as skeletal muscle mass, body fat mass, total body water, and visceral fat area.
Body composition: Body fat (%) | baseline, 12 weeks
  The InBody device is a bioelectrical impedance analysis (BIA) system designed to assess body composition in a non-invasive, rapid, and reliable manner. It quantifies key components such as skeletal muscle mass, body fat mass, total body water, and visceral fat area.
Body composition: Lean mass weight (kg) | baseline, 12 weeks
  The InBody device is a bioelectrical impedance analysis (BIA) system designed to assess body composition in a non-invasive, rapid, and reliable manner. It quantifies key components such as skeletal muscle mass, body fat mass, total body water, and visceral fat area.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No